CLINICAL TRIAL: NCT06942832
Title: The Integration of SPOZ Technology to Support and Enhance the Vitality Acupunch Exercise Program for Improving the Disease Dysfunction and Functional Fitness Deterioration of Older Adults With Dementia
Brief Title: Integrating SPOZ Technology to Support and Enhance the Vitality Acupunch (VA) Exercise Program for Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20240009(2)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Disease and Dysfunction; Functional Fitness Deterioration; Activities of Daily Living; Instrumental Activities of Daily Living; Sleep Quality
MeSH Terms: conditions — Disease; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-SPOZ exercise program (Experimental): The VA-SPOZ exercise program was comprised of 3 parts: (1) the first part had 5 movements, including breathing regulation, alternating arm stretching, trunk movement, alternating left and right legs, and gradually started the blood circulation in a gentle way; (2) the second part had 14 movements, using five punching techniques, the left and right arms alternating in a natural parabola, and punching the acupoints to vibrate meridians. The purpose of the second part of the movement was to stimulate the 14 meridians and to promote the circulation of qi and blood throughout the body; (3) the third part had 5 movements, which were to adjust the breath, relax the muscles, stretch the body, and warm the face and lower back of the body by hand touch. Participants wore SPOZ devices on both hands to record and track the accuracy of the movements.The 40-minute program was administered three times a week for 6 months.
  Interventions: Other: VA-SPOZ exercise program
- Control (Active Comparator): Participants in the control group maintained their routine activities.
  Interventions: Other: Control

INTERVENTIONS:
Other: VA-SPOZ exercise program — The VA-SPOZ exercise program had 3 phases and took 40 minutes to complete. The program was performed in a seated position, and the participants wore SPOZ devices on both hands to record and track the accuracy of the movements.
  Arms: VA-SPOZ exercise program
Other: Control — Participants maintained their routine activities.
  Arms: Control

SUMMARY:
This project was aimed to examine the effects of a six-month VA exercise program incorporated the SPOZ technology in improving the disease dysfunction and functional fitness deterioration of older adults with dementia in adult daycare centers.

DETAILED DESCRIPTION:
A cluster-randomized controlled trial was conducted to examine the effects of a six-month VA exercise program incorporated the SPOZ technology in improving the disease dysfunction, functional fitness deterioration (balance, lower muscle endurance, gait speed, handgrip strength, cardiorespiratory endurance, muscle endurance, agility, body flexibility), activities of daily living, instrumental activities of daily living, and sleep quality of older adults with dementia in adult daycare centers. Using convenience sampling, 10 adult daycare centers with 142 older adults were recruited, and then cluster-randomized by the daycare centers to an experimental or a control group. The experimental group received a 40-minute program 3 times a week for 6 months; the control group maintained their routine activities. The two groups were measured at three time points: before the intervention, and at three months and six months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as dementia by a physician, or
* screened by the SPMSQ as dementia
* age 65 and older

Exclusion Criteria:

* have severe cardiopulmonary disease
* have physical mobility impairment
* have spinal cord injury

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Balance | 6 months
  measured by the Balance tests in SPPB
Lower muscle endurance | 6 months
  measured by the 5-time sit-to-stand in SPPB
Gait speed | 6 months
  measured by the 4-m walk in SPPB
Handgrip strength | 6 months
  measured by the Digital Handgrip Dynamometer (TKK-5101)
Cardiorespiratory endurance | 6 months
  measured by the 2-minute step test
Muscle endurance | 6 months
  measured by the SPOZ devices
Agility | 6 months
  measured by the SPOZ devices
Body flexibility | 6 months
  measured by the SPOZ devices

SECONDARY OUTCOMES:
Activities of daily living (ADL) | 6 months
  measured by the Disability Assessment for Dementia (Categories 1-4). The scale has 47 questions measuring 11 types of activities; of which, 22 questions measuring 4 types of ADL. The scoring system (yes = 1, no = 0, and not applicable = N/A) can be divided into three parts: (1) initiation (7 items): measuring the ability to decide or to start an action; (2) planning and organization (8 items): measuring the ability to structure activities in an appropriate sequence and to be able to prepare relevant supplies or develop strategies before action; and (3) performance (7 items): measuring the ability to complete the entire activity. Divide the total score by the number of questions answered (excluding the number of questions that are not applicable), the score converts into a percentage. A higher percentage indicates less disability in daily activities.
Instrumental activities of daily living (IADL) | 6 months
  measured by the Disability Assessment for Dementia (Categories 5-10). The scale has 47 questions measuring 11 types of activities; of which, 22 questions measuring 6 types of IADL. The scoring system (yes = 1, no = 0, and not applicable = N/A) can be divided into three parts: (1) initiation (6 items): measuring the ability to decide or to start an action; (2) planning and organization (6 items): measuring the ability to structure activities in an appropriate sequence and to be able to prepare relevant supplies or develop strategies before action; and (3) performance (10 items): measuring the ability to complete the entire activity. Divide the total score by the number of questions answered (excluding the number of questions that are not applicable), the score converts into a percentage. A higher percentage indicates less disability in daily activities.
Sleep quality | 6 months
  measured by the Neuropsychiatric Inventory Questionnaire (Item 11). The item 11 measures sleep/nighttime behaviors. The assessment consists of three parts: (1) to determine the presence or absence of symptoms, 0 = no, 1 = yes; (2) to determine the severity of the symptoms, rating between 1 and 3, and with higher scores indicate more severe symptoms; (3) to rate the degree of caregiver's distress caused by the client's symptoms on a scale of 0-5, and with higher scores indicating greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No